CLINICAL TRIAL: NCT03429140
Title: Early Anti-inflammatory Treatment in Patients With Acute ACL Tear and Painful Effusions
Acronym: HEALR
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cale Jacobs, PhD (Other)
Responsible Party: Sponsor-Investigator, Cale Jacobs, PhD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-0662-F6A
Record Dates: First submitted 2017-02-06; First posted 2018-02-12 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Anterior Cruciate Ligament
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Once it has been determined that a subject meets the entry requirements of the study they will be randomized, like the flipping of coin into one of two treatment groups. Neither the subject nor the investigator will be told which of the two treatments that the subject is assigned to. However, the investigator can find out in the case of emergency. Treatment assignment will be released to the subject after they have completed all study visits.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - Gel-One (Experimental): Gel-One (3ml/30 mg Hyaluronan) one time injection at visit 3
  Interventions: Drug: Gel-One
- Group 1 - Saline Placebo (Placebo Comparator): 3 ml saline placebo one time injection at visit 3
  Interventions: Other: Saline Placebo

INTERVENTIONS:
Drug: Gel-One — an injection of Gel-One® (hyaluronan, 3 mL) 1-2 weeks after ACL surgery
  Arms: Group 1 - Gel-One
Other: Saline Placebo — a placebo injection (saline, 3 mL) 1-2 weeks after ACL surgery
  Arms: Group 1 - Saline Placebo

SUMMARY:
This research study is designed to allow the investigator to answer many questions about the reasons why anterior cruciate ligament (ACL) injury leads to knee pain and disability and osteoarthritis.

The purpose of this research is to gather information on how safe and effective Gel-One is in alleviating knee pain following ACL surgery.

DETAILED DESCRIPTION:
This is a single-center, placebo-controlled, double-blinded, randomized controlled trial.

This trial will be conducted at the University of Kentucky's Orthopaedic and Sports Medicine Center (Turfland Facility), with subjects being recruited from the patient populations of UK's Sports Medicine surgeons (Drs. Christian Lattermann, Darren Johnson, Mary Lloyd Ireland, and Scott Mair) during regularly schedule office visits.

After providing informed consent, subjects will be randomized into one of two groups, and there will be 19 subjects per group. All groups will receive standard of care aspiration and triamcinolone injection (40mg, Kenalog) within 1-10 days after ACL injury. The subjects will undergo initial standard of care pre-habilitation as deemed necessary by the surgeon and will undergo ACL reconstruction surgery. Knee aspiration will be performed 7-10 days after ACL reconstruction surgery and the patients will be randomized into 1 of 2 groups:

* Group 1: will receive injection of Gel-One (3ml 30mg Hyaluronan)
* Group 2: will receive an injection of 3ml of a saline placebo

Knee Aspiration: All subjects will undergo a total of four aspirations.

Visit Schedule and Procedures:

Visit 1 Screening (1-10 days post injury): Upon arriving at the clinic potential subjects will have the following assessments: range of motion, knee instability (Lachman's test) and standardized Flexion weight bearing x-rays, all of which are the standard of care for a patient with a suspected ACL injury. After providing informed consent to participate in the study, subjects will be asked to fill in standard questionnaires.

Collection of urine and 10 cc of blood for laboratory testing, partial Medical history, concomitant medications, demographic information, body mass index (BMI) measurement, smoking status, and questions will be collected. Scheduling for study-related magnet resonance imaging (MRI) scans.

Visit 2 (day of surgery)

* Lab specimens collected (urine and 10cc of blood)
* Pain Questionnaires administered prior to surgery
* Knee aspiration (in the operating room under anesthesia, both knees)
* Patient reported outcomes (PROs) administered prior to surgery

Visit 3 (1-2 weeks post surgery)

* Pain Questionnaires administered
* Lab tests (urine and 10cc of blood)
* Randomization into group 1 or 2
* Knee aspiration and administration of either 3ml of saline(placebo) or Hyaluronan (study drug)

Visit 4 (4-6 weeks post surgery)

* Pain Questionnaire administered
* Knee aspiration and lab specimens collected
* Patient reported outcomes (PROs) administered

Visit 5 (6 months follow-up/Early Termination Visit)

* Patient reported outcomes (PROs) administered
* Pain Questionnaires administered
* Functional laboratory testing

Visit 6 (12 months follow-up/Early Termination Visit)

* Patient reported outcomes (PROs) administered
* Pain Questionnaires administered
* Functional laboratory testing
* MRI scan

There are no costs associated with either the study medications and study-specific laboratory and imaging analyses. Either the participant or their insurance company, Medicare or Medicaid will be responsible for the costs of all care and treatment a participant receives during this study that they would normally receive for their condition. These are costs that are considered medically reasonable and necessary and will be part of the care a patient would receive if they did not take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* 14-33 years of age
* Currently participating in a sporting activity
* ACL injury occurred while playing in a sporting activity
* Normal contralateral knee status
* Documentation of closed growth plates as noted on the screening x-rays

Exclusion Criteria:

* Underlying inflammatory disease (i.e. Rheumatoid Arthritis, Psoriatic Arthritis etc)
* Currently have any infections, including infection of the skin, or have signs and symptoms of an infection, including fever
* Have a disease that weakens your immune system such as diabetes, cancer, HIV or AIDs
* Other major medical condition requiring treatment with immunosuppressant or modulating drugs
* A history of chronic use of non-steroidal anti-inflammatory drugs
* Received corticosteroid injections into the injured knee within three months of enrollment
* History of allergic reaction to hyaluronan injections
* Previous exposure or allergic reaction to Kenalog®
* Prior knee surgery (Ipsilateral or contralateral)
* Have received any investigational drug with 4 weeks of study Visit 1

Ages: 14 Years to 33 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2019-06-23 (Actual); Study Completion 2019-06-23 (Actual)

PRIMARY OUTCOMES:
Change in KOOS score over time | 12 months
  Knee Injury and Osteoarthritis Outcome Score (KOOS) symptoms

SECONDARY OUTCOMES:
Change in CTX-II pre and post surgery | up to 4 weeks
  CTX -II ELISA measurements

OTHER OUTCOMES:
MRIT1rho measurement of articular cartilage | 12 months
  MRI measurement
Number of participants with adverse events that are related to treatment. | 12 months
  Protocol safety questionnaires and SAE/AE reporting

CONTACTS AND LOCATIONS:
Overall Officials: Cale Jacobs, PhD, Principal Investigator — University of Kentucky
Locations (1):
- UK Healthcare at Turfland, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No